CLINICAL TRIAL: NCT04198025
Title: Evaluating the Association Between Psoas Density Measurement on Preoperative CT Imaging and Postoperative Outcomes
Brief Title: Psoas Density in Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: Psoas Muscle Density
Record Dates: First submitted 2019-11-19; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-10

CONDITIONS: Cancer of Colon
Keywords: psoas muscle density; frailty
MeSH Terms: conditions — Colonic Neoplasms; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent colorectal resection: Patients in this observational study will have undergone CT scan as routine work up prior to resection of elective colorectal cancer.
  Psoas muscle density will be measured (in Hounsfield units from CT images) at lumbar vertebral level L3.

SUMMARY:
Colorectal cancer (CRC) is the 3rd most common cancer worldwide. In the UK, CRC is the 4th most common cancer accounting for 12% of cancers diagnosed each year with approximately 41,300 new cases diagnosed in 2014. Surgery remains the only treatment option that can reliably achieve cure from colorectal cancer and thus nearly 20,000 major bowel resections are performed for this yearly in the UK. Surgery for these cancers however carries risk of major complications and potentially death. Selecting appropriate patients for surgery remains a challenge to cancer teams.

Risk factors exist for complications after surgery for CRC, many of which can be assessed and discussed with the patient prior to surgery, so that any decision to operate is with fully informed consent from the patient. Increasing attention is being paid to a patient's frailty or fitness as one of these risk factors. Our centre has previously shown that measuring the cross-sectional area of the psoas muscle (a large muscle near the spine) from preoperative imaging could predict major complications in colorectal cancer patients (Jones 2015), however specialist software and patient height is required to make this calculation. More recently we have demonstrated that the measurement of the psoas muscle density on preoperative imaging (i.e. routine CT scans that all patients have before surgery to plan treatment), may potentially be useful to predict which patients are at most risk of a major complication (Herrod 2019). If this finding holds true when tested on a larger scale, it could be used to help surgical teams make the decision on whether to offer surgical resection, what kind of operations to perform, how to best support individuals undergoing operation and to ensure that the patient has the most information available to decide what risk they are at by having major surgery.

ELIGIBILITY:
Inclusion Criteria:

Patient criteria:

* Having a major colorectal resection for the treatment of cancer
* Elective or emergency surgery
* Adults, defined as age ≥18 years of age (no maximum limit)
* Had a preoperative CT scan of the abdomen with contrast (portal venous phase)
* Operation performed between 31st Aug 2013 - 31st Aug 2019

Exclusion Criteria:

* Not having a preoperative CT scan with contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective analysis of patients (>18 years old) having undergone curative colorectal resection for cancer (between 31st Aug 2013 - 31st Aug 2019) in one if this multicentre study sites. All patients must have undergone preoperative CT scan with contrast.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of post operative complications (Clavien-Dindo grade 3-4) during inpatient hospital stay. | Through study completion, an average of 10 days.
  Recorded post operative complications requiring intervention during post operative stay until initial discharge from hospital.

SECONDARY OUTCOMES:
Post operative length of stay | Through study completion, usually between 6-10 days.
  Number of days
Mortality | Up to 5 year follow up from operation
  Recorded patient death
Post operative complications beyond hospital discharge. | From hospital discharge to record review (i.e. 30 days, 90 days, 2 - 5 year follow up).
  Recorded post operative complications (including re-operation or recurrence) until discharge from surgical clinic or date of record review.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Graduate Entry Medicine, Royal Derby Hospital, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No